CLINICAL TRIAL: NCT01828710
Title: Effect of Treatment With Myo-inositol on Human Semen Parameters in Patients Undergoing IVF Cycles
Brief Title: Myo-inositol on Human Semen Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AGUNCO Obstetrics and Gynecology Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: INO-2103-GC
Record Dates: First submitted 2013-03-21; First posted 2013-04-11 (Estimated); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Asthenozoospermia; Oligospermia
Keywords: Myo-inositol; oligoasthenoteratospermia; semen parameters; IVF
MeSH Terms: conditions — Asthenozoospermia; Oligospermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Myo-inositol normospermic (Sham Comparator): 29 normospermic treated with 4000mg/die of myo-inositol and 400 µg of folic acid
  Interventions: Dietary Supplement: Myo-inositol normospermic
- Myo-inositol OAT (Active Comparator): 13 OAT patients treated with 4000mg/die of myo-inositol associated to 400 µg of folic acid
  Interventions: Dietary Supplement: Myo-inositol OAT
- Folic acid normospermic (Placebo Comparator): 20 normospermic patients treated with 400 µg of folic acid
  Interventions: Dietary Supplement: Folic Acid normospermic

INTERVENTIONS:
Dietary Supplement: Myo-inositol normospermic — 4000mg/die of myo-inositol and 400 µg of folic acid (Inofolic® Lo.Li. pharma s.r.l., Roma) for three months.
  Arms: Myo-inositol normospermic
Dietary Supplement: Myo-inositol OAT — B 13 OAT patients treated with 4000mg/die of myo-inositol associated to 400 µg of folic acid (Inofolic® Lo.Li. pharma s.r.l., Roma) for three months
  Arms: Myo-inositol OAT
Dietary Supplement: Folic Acid normospermic — Group C 20 normospermic patients treated with 400 µg of folic acid (kindly provided by Lo.Li. pharma s.r.l., Roma) for three months.
  Arms: Folic acid normospermic

SUMMARY:
Many clinical evidences suggest that Myo-inositol plays a crucial role in human reproduction. Also, it was shown that Myo-inositol concentration in the seminiferous tubules was higher than in serum, and interestingly it was increasing through the epididymis and the deferent duct mining that sperm cell before ejaculation are stored in a "medium" highly enriched in myo-inositol.

Starting from this evidences, the investigators hypothesized that myo-inositol may be a possible factor able to improve the semen parameters of samples used in in vitro fertilization cycles.

DETAILED DESCRIPTION:
Samples of seminal fluid were obtained from two groups of patients undergoing to an IVF cycle: healthy normospermic subjects and subjects with oligoasthenoteratospermia (OAT, < 15 mil/ml).

Semen volume, spermatozoa number and motility were evaluated during the initial semen analysis and after density gradient separation method. These parameters were evaluated before and after the administration of 4000mg/die of myo-inositol associated to 400 µg of folic acid (Inofolic lolipharma Rome) for three months.

A third group of healthy normospermic subject were traded with 400 µg of folic acid for three months and was consider a control group.

ELIGIBILITY:
Inclusion Criteria:

Undergoing to IVF cycle OAT

Exclusion Criteria:

No undergoing to IVF cycle

Ages: 25 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2012-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
sperm concentration | after 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Marco Palumbo, M.D., Principal Investigator — University of Catania - Department of Surgery - Section of Obstetrics and Gynecology - Centre of Physiopathology of Reproduction; Gianfranco Carlomagno, Ph.D., Study Director — A.G.Un.Co. Obstetrics and gynaecology center
Locations (1):
- Centre of Physiopathology of Reproduction, Catania, CT, Italy

REFERENCES:
- [Derived] de Ligny W, Smits RM, Mackenzie-Proctor R, Jordan V, Fleischer K, de Bruin JP, Showell MG. Antioxidants for male subfertility. Cochrane Database Syst Rev. 2022 May 4;5(5):CD007411. doi: 10.1002/14651858.CD007411.pub5. PMID 35506389